CLINICAL TRIAL: NCT01370369
Title: A Phase 2 Open-Label, Sequential Dose Escalation Study to Evaluate the Efficacy, Pharmacokinetics and Safety of Three Volumes (1.25, 2.50 and 3.75 mL) of Testosterone Gel 2% (FE 999303) Equivalent to 23, 46 And 70 mg of Testosterone in Hypogonadal Males
Brief Title: Efficacy, Pharmacokinetics and Safety of Testosterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000011
Record Dates: First submitted 2011-06-01; First posted 2011-06-09 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Testicular Hypogonadism
MeSH Terms: conditions — Eunuchism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Single Testosterone Dose (Inner Thigh) (Experimental): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the inner thigh followed by a seven day washout period.
  Interventions: Drug: Testosterone gel (FE 99903)
- Single Testosterone Dose (Abdomen) (Experimental): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the abdomen followed by a seven day washout period.
  Interventions: Drug: Testosterone gel (FE 99903)
- Single Testosterone Dose (shoulder/upper arm) (Experimental): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the shoulder/upper arm.
  Interventions: Drug: Testosterone gel (FE 99903)
- Testosterone 1.25 (Experimental): Subjects received testosterone gel 2% at dose of 1.25 mL (one stroke) applied once daily for 10 consecutive days to the shoulder/upper arm.
  Interventions: Drug: Testosterone gel (FE 99903)
- Testosterone 2.50 (Experimental): Subjects received testosterone gel 2% at dose of 2.50 mL (two strokes) applied once daily for 10 consecutive days to the shoulder/upper arm.
  Interventions: Drug: Testosterone gel (FE 99903)
- Testosterone 3.75 (Experimental): Subjects received testosterone gel 2% at dose of 3.75 mL (three strokes) applied once daily for 10 consecutive days to the shoulder/upper arm.
  Interventions: Drug: Testosterone gel (FE 99903)

INTERVENTIONS:
Drug: Testosterone gel (FE 99903)

SUMMARY:
This is an open-label study of a single and repeated application of three dose levels of topical testosterone in hypogonadal males with morning serum testosterone concentrations < 297 ng/dL.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* History of hypogonadism
* In good health based on medical history, physical examination and clinical laboratory tests
* Screening morning serum testosterone ≤ 297 ng/dL
* One or more symptoms of testosterone deficiency (i.e. fatigue, reduced libido or reduced sexual functioning of non-vasculogenic or neurogenic nature)
* Body mass index (BMI) between 18 and 31

Exclusion Criteria:

* Prostate cancer
* Palpable prostatic mass(es)
* Generalized skin irritation or significant skin disease
* Use of any medications that could be considered anabolic (e.g. dehydroepiandrosterone (DHEA)) or could interfere with androgen metabolism (e.g. spironolactone, finasteride, ketoconazole)
* Clinically significant anemia or renal dysfunction
* Hyperparathyroidism or uncontrolled diabetes
* Serum PSA Levels; ≥ 4ng/mL
* History of cardiovascular disease
* Use of estrogens, Gonadotropin-releasing hormone (GnRH) agonists/antagonist, human growth hormone (hGH), (within previous 12 months)
* Use of testosterone products (within eight months for parenteral products, or six weeks for other preparations)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- AccuMed Research Associates, Garden City, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one study site in the US. Out of 42 subjects screened, 20 subjects were enrolled in the study.
Pre-assignment Details: Apart from having history of hypogonadism, the study subjects were required to present with one or more symptoms of low testosterone (i.e. fatigue, decreased muscle mass, reduced libido, reduced sexual functioning of a non-mechanical nature). The study subjects needed to be in good health despite exhibiting hypogonadism.
Groups:
- Testosterone Topical: For single dose pharmacokinetics (PKs), a single application of 2.50 mL (two strokes) of the testosterone gel 2% was applied to the inner thigh followed by a 7-day washout period. After this washout period, the second single application of 2.50 mL (two strokes) of the testosterone gel 2% was applied to the abdomen followed by another 7-day washout period. After this washout period, the third single application of 2.50 mL (two strokes) of the testosterone gel 2% was applied to the shoulder/upper arm.
  After the last 24 hour PK sampling from the shoulder/upper arm, three ascending doses of testosterone gel 2%, 1.25, 2.50 and 3.75 mL (one stroke, two strokes and three strokes, respectively), were sequentially applied once daily for 10 consecutive days to the shoulder/upper arm. Steady-state PK evaluations were performed starting on the morning of the last administered dose. There was no washout between each of the 10-day treatments.
Period: Overall Study
Arm/Group | Testosterone Topical
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The data are presented for Intent-to-treat (ITT) population, which comprised of all subjects who received at least one dose of the Investigational Medicinal Product (IMP). In this study, the safety, ITT, full analysis set (FAS) and per protocol (PP) populations were identical.
Groups:
- Testosterone Topical: For single dose PKs, a single application of 2.50 mL (two strokes) of the testosterone gel 2% was applied to the inner thigh followed by a 7-day washout period. After this washout period, the second single application of 2.50 mL (two strokes) of the testosterone gel 2% was applied to the abdomen followed by another 7-day washout period. After this washout period, the third single application of 2.50 mL (2 strokes) of the testosterone gel 2% was applied to the shoulder/upper arm.
  After the last 24 hour PK sampling from the shoulder/upper arm, 3 ascending doses of testosterone gel 2%, 1.25, 2.50 and 3.75 mL (1 stroke, 2 strokes and 3 strokes, respectively), were sequentially applied once daily for 10 consecutive days to the shoulder/upper arm. Steady-state PK evaluations were performed starting on the morning of the last administered dose. There was no washout between each of the 10-day treatments.
Arm/Group | Testosterone Topical
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: year] | 47.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 28.3 (2.3)
Height [Mean (Standard Deviation); unit: Inch] | 69.7 (3.2)
Weight [Mean (Standard Deviation); unit: lbs] | 196.2 (23.3)

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate - the Percentage of Subjects Whose Minimum Concentration Observed (Cmin) and Average Steady State Concentration (Cave) of Serum Testosterone Levels Were Between 298 and 1043 ng/dL.
Description: Responder rate was calculated for the subjects who received 10 days of treatment with three doses of testosterone gel; 1.25 mL, 2.50 mL, and 3.75 mL, respectively. The data were presented using descriptive statistics for this outcome.
Time Frame: From Baseline to Day 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Number; unit: percentage of subjects
Groups:
- Testosterone 1.25: Subjects received testosterone gel 2% at dose of 1.25 mL (one stroke - equivalent to 23 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
- Testosterone 2.50: Subjects received testosterone gel 2% at dose of 2.50 mL (two strokes - equivalent to 46 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
- Testosterone 3.75: Subjects received testosterone gel 2% at dose of 3.75 mL (three strokes - equivalent to 70 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
percentage of subjects
  Cave | 73.7 | 77.7 | 75.0
  Cmin | 20.0 | 40.0 | 55.0

2. Secondary Outcome: Pharmacokinetic Parameter : Maximum Concentration Observed (Cmax) for Total Testosterone, After an Initial Single Treatment (Testosterone) on the Abdomen, Inner Thigh and Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 1, 7 and 13
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Single Testosterone Dose (Inner Thigh): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the inner thigh followed by a 7-day washout period.
- Single Testosterone Dose (Abdomen): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the abdomen followed by a 7-day washout period.
Arm/Group | Single Testosterone Dose (Inner Thigh) | Single Testosterone Dose (Abdomen) | Single Testosterone Dose (Shoulder/Upper Arm)
Number analyzed (Participants) | 20 | 20 | 20
ng/dL | 519 (171) | 451 (157) | 926 (737)

3. Secondary Outcome: Pharmacokinetic Parameter : Time of Maximum Observed Concentration (Tmax) for Total Testosterone, After an Initial Single Treatment (Testosterone) on the Abdomen, Inner Thigh, and Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 1, 7 and 13
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Median (Full Range); unit: hour
Groups:
- Single Testosterone Dose (Abdomen): Subjects received a single application of 2.50 mL (two strokes) of the testosterone gel 2% applied to the abdomen thigh followed by a seven day washout period.
Arm/Group | Single Testosterone Dose (Inner Thigh) | Single Testosterone Dose (Abdomen) | Single Testosterone Dose (Shoulder/Upper Arm)
Number analyzed (Participants) | 20 | 20 | 20
hour | 24.0 [0.0 to 24.8] | 9.0 [2.0 to 24.0] | 11.0 [4.0 to 24.7]

4. Secondary Outcome: Pharmacokinetic Parameter : Area Under the Plasma Concentration Time Curve From 0 to 24 hr (AUC0-24) Observed for Total Testosterone, After an Initial Single Treatment (Testosterone) on the Abdomen, Inner Thigh and Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 1, 7 and 13
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP. Number of subjects was less than 20 in some group(s) for AUC0-24 as parameter could not be calculated due to missing concentration for 0 hr.
Measure: Mean (Standard Deviation); unit: ng*hour/dL
Arm/Group | Single Testosterone Dose (Inner Thigh) | Single Testosterone Dose (Abdomen) | Single Testosterone Dose (Shoulder/Upper Arm)
Number analyzed (Participants) | 20 | 19 | 20
ng*hour/dL | 9472 (2306) | 8918 (2924) | 13368 (7163)

5. Secondary Outcome: Pharmacokinetic Parameter - Cmax for Total Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
ng/dL | 586 (290) | 907 (783) | 1258 (774)

6. Secondary Outcome: Pharmacokinetic Parameter - Tmax for Total Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
hour | 6.0 [0.0 to 24.0] | 4.0 [0.0 to 24.9] | 6.0 [0.0 to 24.0]

7. Secondary Outcome: Pharmacokinetic Parameter : AUC0-24 Observed for Total Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP. Number of subjects was less than 20 in some group(s) for AUC0-24 as parameter could not be calculated due to missing concentration for 0 and/or 24 hr.
Measure: Mean (Standard Deviation); unit: ng*hour/dL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 19 | 18 | 20
ng*hour/dL | 9229 (2946) | 12148 (6300) | 17625 (9250)

8. Secondary Outcome: Pharmacokinetic Parameter - Cmax for Free Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
pg/mL | 134 (90) | 229 (273) | 382 (342)

9. Secondary Outcome: Pharmacokinetic Parameter - Tmax for Free Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
hour | 6.0 [0.0 to 24.3] | 7.0 [0.0 to 24.9] | 6.0 [0.0 to 24.0]

10. Secondary Outcome: Pharmacokinetic Parameter : AUC0-24 Observed for Free Testosterone With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg*hour/mL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 18 | 14 | 17
pg*hour/mL | 1765 (781) | 2655 (2078) | 4663 (3517)

11. Secondary Outcome: Pharmacokinetic Parameter - Cmax for Dihydrotestosterone (DHT) With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
ng/dL | 64.4 (32.2) | 93.3 (51.9) | 120 (60)

12. Secondary Outcome: Pharmacokinetic Parameter - Tmax for DHT With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: ITT population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Median (Full Range); unit: hour
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
hour | 6.0 [0.0 to 24.4] | 4.0 [0.0 to 24.9] | 6.0 [0.0 to 25.0]

13. Secondary Outcome: Pharmacokinetic Parameter : AUC0-24 Observed for DHT With Multiple-dose Profile of IMP After 10 Days of Treatment to Shoulder/Upper Arm.
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: Samples were collected at pre-dose and at 2, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 23, 33, and 43
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*hour/dL
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 14 | 16 | 18
ng*hour/dL | 1063 (479) | 1458 (726) | 1974 (890)

14. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: The data were presented using descriptive statistics for this outcome.
Time Frame: From Baseline to Day 43
Population: Safety Analysis Set population was used for this analysis, which comprised of all subjects who received at least one dose of the IMP.
Measure: Number; unit: number of event
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Number analyzed (Participants) | 20 | 20 | 20
number of event | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Overall Treatment Period (43 days)
Description: The treatment-emergent adverse event (TEAE), defined as any AE occurring after start of IMP administration and within the time of residual drug effect (5 days) (including PK assessment periods), or a pretreatment AE or preexisting medical condition that worsens in intensity after start of IMP, were presented.
Groups:
- Testosterone 1.25: Subjects received testosterone gel 2% at dose of 1.25 mL (1 stroke - equivalent to 23 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
- Testosterone 2.50: Subjects received testosterone gel 2% at dose of 2.50 mL (2 strokes - equivalent to 46 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
- Testosterone 3.75: Subjects received testosterone gel 2% at dose of 3.75 mL (3 strokes - equivalent to 70 mg of testosterone) applied once daily for 10 consecutive days to the shoulder/upper arm.
Arm/Group | Testosterone 1.25 | Testosterone 2.50 | Testosterone 3.75
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone 1.25 (N=20) | Testosterone 2.50 (N=20) | Testosterone 3.75 (N=20)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 2
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a restriction on joint publications prepared in collaboration between investigator and sponsor as Ferring reserves the right to be involved in this decision. In the event of any disagreement in the content of any publication both investigator's and Ferring´s opinion will be fairly and sufficiently represented in the publication.